CLINICAL TRIAL: NCT06068829
Title: A Multicentric, Retrospective, Real-Word Study to Evaluate the Efficacy and Safety of Inebilizumab Compare With Rituximab in Neuromyelitis Optica Spectrum Disorders
Brief Title: Inebilizumab and Rituximab in Neuromyelitis Optica Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Feng Jinzhou (Other)
Responsible Party: Sponsor-Investigator, Feng Jinzhou, Ph.D, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: IRNMO-001
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
Keywords: Neuromyelitis Optica Spectrum Disorders; Inebilizumab; Rituximab
MeSH Terms: conditions — Neuromyelitis Optica | interventions — inebilizumab; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples are collected before the treatment and at the last follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group 1: Intravenous methylprednisolone (IVMP) plus Inebilizumab
  Interventions: Drug: Inebilizumab
- Exposed group 2: IVMP plus Rituximab (RTX)
  Interventions: Drug: Rituximab(RTX)

INTERVENTIONS:
Drug: Inebilizumab — Inebilizumab: 300mg IV on Day1 and Day 15. The first dose of inebilizumab was given after IVMP.
  Groups: Exposed group 1
Drug: Rituximab(RTX) — RTX: 500mg IV on Day 1 and Day15. The first dose of RTX was given after IVMP.
  Groups: Exposed group 2

SUMMARY:
To compare the safety and efficacy of Inebilizumab and Rituximab in neuromyelitis optica spectrum disorders (NMOSD) patients.

DETAILED DESCRIPTION:
Inebilizumab is a humanized anti-CD19 monoclonal antibody. CD19 is broadly expressed on B-lineage cells, particularly late-stage memory B-lymphocytes and plasma blasts. Inebilizumab depletes antibody-secreting plasmablasts and some plasma cells.

Rituximab (RTX) is a chimeric anti-CD20 monoclonal antibody that promotes B-lymphocyte depletion through antibody-dependent cellular cytotoxicity (ADCC)/complement-dependent cytotoxicity (CDC), promotes an immunoregulatory T-lymphocyte phenotype, and activates neutrophil/macrophage phagocytosis.

This is a retrospective, multicentre, real-world study which aims to compare Inebilizumab with RTX in neuromyelitis optica spectrum disorders patients. Eighty patients from 8 centres in China will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years with anti-AQP4-IgG seropositive NMOSD as defined by 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).
* 2. Expanded disability status scale (EDSS) score ≤ 8 and ≥ 2.5 during the acute phase.
* 3. Patients have given their written informed consent.

Exclusion Criteria:

* 1. Lactating and pregnant females.
* 2. Participate in other interventional studies within 30 days or within 5 half-lives of the investigational agent before received inebilizumab and rituximab (RTX).
* 3. Receipt of any experimental B-cell depleting agent within 6 months prior inebilizumab and RTX, and B-cells below the lower limit of normal
* 4. Known history of a severe allergy or reaction to any component of the investigational product formulation.
* 5. Known active severe bacterial, viral, or other infection or any major episode of infection requiring hospitalization (including viral hepatitis, active tuberculosis or positive tuberculosis screening).
* 6. History of alcohol, drug, or chemical abuse, or a recent history of such abuse < 1 year prior to treatment.
* 7. History of malignancies.
* 8. Combined with severe mental disorders and other conditions and unable to cooperate with follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Neuromyelitis Optica Spectrum Disorders
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale Score (EDSS) from baseline. | 12 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline to 12 months after treatment (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Time to first relapse | 12 months
  Relapse: A monophasic clinical episode with patient-reported symptoms and objective findings reflecting a focal or multifocal inflammatory demyelinating event in the central nervous system (CNS), developing acutely or subacutely, with a duration of at least 24h, without fever or infection.
Number of new, and/or enlarging T2- hyperintense lesions detected by Magnetic Resonance Imaging (MRI) | 12 months
  Number of new, and/or enlarging T2-hyperintense lesions detected by Magnetic Resonance Imaging (MRI) at the last visit.

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline | 6 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline at month 6 (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Percentage of Participants with Disability Improvement | 12 months
  Disability improvement is defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5(EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Percentage of Participants with Disability Worsening | 12 months
  A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
Change in modified Rankin score (mRS) from baseline | 12 months
  Change in modified Rankin score (mRS) from baseline at month 12(mRS: Minimum Score 0, Maximum score 6, higher scores mean a worse outcome).
Change in Timed 25 Foot Walk Test from baseline | 12 months
  Change in time taken to complete the timed 25foot walk test from baseline
Number of NMOSD attacked related rescue treatment. | 12 months
Annual relapse rate (ARR) before and after Inebilizumab/Rituximab | 12 months
  ARR will be measured in the baseline (according to patients' history before inebilizumab/rituximab) and after 12 months of intervention.
Change in serum glial fibrillary acidic protein antibody (GFAP-Ab) levels from baseline. | 12 months
  Change in serum GFAP-Ab levels from baseline at the last visit
Change in aquaporin 4 antibody (AQP4-Ab) titers from baseline. | 12 months
  Change in AQP4-ab titers from baseline at the last visit.
Change in serum Neurofilament light chain protein (NfL) levels from baseline. | 12 months
  Change in serum NfL levels from baseline at the last visit.
Change in Visual Acuity (VA) from baseline | 12 months
  Change in Visual Acuity (VA) at month 12.
Changes in The Five Level of EuroQol Five Dimensions Questionnaire (EQ-5D-5L) scores from baseline | 12 months
  Changes in EQ-5D scores from baseline at month 12(EQ-5D-5L: Minimum Score 5, Maximum score 25, lower scores mean a better quality of life).
Change in retinal nerve fiber layer (RNFL) loss from baseline | 12 months
  Change in retinal nerve fiber layer (RNFL) loss measured by optical coherence tomography (OCT) from baseline at month 12.
Adverse reactions during treatment and follow-up | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Feng, Ph.D, Principal Investigator — First Affiliated Hospital of Chongqing Medical University